# **COVER PAGE**

OFFICIAL TITLE

The Effect of Digital Interactive and Face-to-Face Peer Support on Medical Students'

NCT NUMBER

not assigned

DOCUMENT TYPE

Informed Consent Form (ICF) - Medical Students

DOCUMENT DATE

16 Sep 2025

UNIQUE PROTOCOL ID

2023-YÖNP-0719

**VERSION** 

v1.0

LANGUAGE

English

#### INFORMED CONSENT FORM

Study Title: The Effect of Digital Interactive and Face-to-Face Peer Support on Medical Students' Clinical Skill Performance, Reflection Skills, and Retention of Clinical Skills

Unique Protocol ID: 2023-YÖNP-0719

Document Date: 16 Sep 2025 — Version: v1.0

#### 1. Introduction

You are invited to take part in a research study conducted by Mustafa Onur YURDAL. Please read this information carefully before deciding whether to participate. If anything is unclear, you may ask questions at any time.

# 2. Purpose of the Study

The purpose of this study is to examine the effects of a digital interactive peer-support program and face-to-face peer support on medical students' clinical skill performance, reflection skills, and retention of clinical skills.

### 3. Procedures and Time Commitment

If you agree to participate, you will be randomly assigned to one of three groups: (1) Digital interactive peer support; (2) Face-to-face peer support; or (3) Standard training (usual curriculum). You will complete learning activities according to your group and complete assessments including an Objective Structured Clinical Examination (OSCE) and a reflection skills questionnaire. The total time commitment is approximately 6 hours.

Approximately 98 participants will take part in this study.

### 4. Risks and Discomforts

This is a minimal-risk educational study. Potential discomforts are limited to the time required for training and assessments, and possible temporary fatigue during practice sessions. No drugs or medical devices are used.

### 5. Benefits

You may or may not benefit directly. Participation may contribute to improved understanding of peer-support approaches in medical education and may help enhance clinical skills training programs.

# 6. Voluntary Participation and Withdrawal

Participation is entirely voluntary. You may refuse to participate or withdraw at any time without penalty or any effect on your grades, standing, or access to educational services.

# 7. Confidentiality

Your information will be kept confidential to the extent permitted by law and institutional policy. Data will be de-identified and stored on secure systems.

Publications or presentations will use aggregate, anonymized data without identifying you.

### 8. Photos and Video

Photos and video recordings may be taken during the study to support educational procedures and quality assurance. If recordings are used for research presentations or publications, faces will be blurred or otherwise de-identified so that participants cannot be recognized. Recordings will not be used in identifiable form without your explicit consent.

## 9. Compensation and Costs

There is no payment for participation and no additional costs to you.

#### 10. Contacts

If you have questions about the study, please contact the research team at the Faculty of Medicine. For questions about your rights as a participant, contact the institutional ethics committee.

#### 11. Consent

By signing below, you acknowledge that you have read and understood the information provided above, had the opportunity to ask questions, and agree to participate voluntarily.

| Participant Name (print): |
|---------------------------|
| Signature: |
| Date: |